CLINICAL TRIAL: NCT04742010
Title: Zoledronic Acid for Prevention of Bone Loss After BAriatric Surgery (ZABAS)
Acronym: ZABAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stinus Gadegaard Hansen (Other)
Collaborators: Research Unit of Health Sciences, Hospital of South West Jutland (Unknown); Department of Regional Health Research, University of Southern Denmark (Unknown); OPEN - Odense Patient data Explorative Network, The University of Southern Denmark, Odense, Denmark (Unknown); Department of Radiology and Nuclear Medicine, Hospital of Southwest Jutland, 6700 Esbjerg, Denmark (Unknown); Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Stinus Gadegaard Hansen, Endocrinologist, Associate professor, PhD, Esbjerg Hospital - University Hospital of Southern Denmark
Organization: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20/41068
Record Dates: First submitted 2021-01-27; First posted 2021-02-05 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Bone Loss; Muscle Atrophy; Bariatric Surgery
MeSH Terms: conditions — Bone Diseases, Metabolic; Muscular Atrophy | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zoledronic Acid (Experimental): Active treatment
  Interventions: Drug: Zoledronic Acid
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic Acid — * A single treatment 21 days before bariatric surgery with Zoledronic acid 5 mg or placebo (an interval of 5 to 180 days is accepted)
  * Pharmaceutical form: Solution for infusion (100 ml normal saline containing 5 mg zoledronic acid or placebo)
  * Administration: slow intravenous infusion with a duration of at least 15 minutes
  Arms: Zoledronic Acid
Drug: Placebo — as above
  Arms: Placebo

SUMMARY:
In a randomised placebo-controlled trial assess effects of zoledronic acid for prevention of bone and muscle loss after bariatric surgery.

DETAILED DESCRIPTION:
In individuals with severe obesity, bariatric surgery effectively reduces body weight, improves obesity related diseases and lowers mortality. A loss of bone and muscle mass and an increase in bone fracture risk are however seen after surgery. In this study it is examined if treatment with zoledronic acid (a drug used to treat osteoporosis) can prevent the bone and muscle loss after bariatric surgery. A single infusion of zoledronic acid or placebo is given before surgery. The study is blinded and randomized for methodological reasons. Bone and muscle scans, tests of muscle strength and physical performance and blood samples (for analysis of markers related to bone and muscle metabolism) are performed at inclusion and 12 and 24 months after surgery. A total of 60 adult individuals will participate. Results will be important for the evidence-based care of patients undergoing bariatric surgery and zoledronic acid.

Study design This is a single center randomized double-blind placebo-controlled study of zoledronic acid for prevention of bone and muscle loss after bariatric surgery. Routine bariatric surgery (RYGB or gastric sleeve) will be performed. The end of study is 24 months after surgery.

Study Population Patients referred for bariatric surgery at The Hospital South West Jutland, Esbjerg will be invited to participate.

Randomization After inclusion and baseline assessment, patients will be randomly assigned to either zoledronic acid or placebo with a 1:1 allocation. A randomization code stratifying an equal number of participants having RYGB or SG into each study arm will be applied.

ELIGIBILITY:
Inclusion Criteria:

* 35 years old or older
* Eligible for bariatric surgery (BMI>35 kg/m2 with obesity-related comorbidity)

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Chronic kidney disease with estimated GFR<45 ml/min.
* Hypocalcemia .
* Hypersensitivity to bisphosphonates, mannitol, sodium citrate or water.
* Metabolic bone disease (osteoporosis is allowed).
* Prior treatment with anti-osteoporotic agents.
* Treatment with oral glucocorticoids
* Other diseases with known effects on bone metabolism

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Quantitative Computed Tomography (QCT) | Change from baseline to 12 and 24 months after bariatric surgery
  Volumetric bone mineral density at the lumbar spine (L1 -L2) (Mindways QCT Pro software, Texas, USA).

SECONDARY OUTCOMES:
QCT | Change from baseline to 12 and 24 months after bariatric surgery
  Volumetric BMD at the proximal femur (Mindways QCT Pro software, Texas, USA).
Biochemical calcium-metabolic markers | Change from baseline to 12 and 24 months after bariatric surgery
  Calcium, parathyroid hormone, vitamin D and markers of bone remodeling (CTX, P1NP).
DEXA | Change from baseline to 12 and 24 months after bariatric surgery
  Bone mineral density at the lumbar spine and total hip (Hologic Discovery, Waltham, MA, US).
HR-pQCT | Change from baseline to 12 and 24 months after bariatric surgery
  Radius and tibia bone microarchitecture (Scanco Medical AG, Brutisellen, Switzerland).
Cortical bone stiffness | Change from baseline to 12 and 24 months after bariatric surgery
  Cortical bone material strength index (BMSi) assessed using microindentation at the anterior surface of the mid-tibia diaphysis (OsteoProbe, Active Life Scientific, California, US).
Muscle Strength | Change from baseline to 12 and 24 months after bariatric surgery
  Upper and lower limb muscle strength assessed using dynamometers (foot, knee, shoulder, hand)
Physical function | Change from baseline to 12 and 24 months after bariatric surgery
  Short physical performance battery (SPPB), Stair Climb, 2 minute walking test

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital South West Jutland, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng M, Fleming T, Robinson M, Thomson B, Graetz N, Margono C, Mullany EC, Biryukov S, Abbafati C, Abera SF, Abraham JP, Abu-Rmeileh NM, Achoki T, AlBuhairan FS, Alemu ZA, Alfonso R, Ali MK, Ali R, Guzman NA, Ammar W, Anwari P, Banerjee A, Barquera S, Basu S, Bennett DA, Bhutta Z, Blore J, Cabral N, Nonato IC, Chang JC, Chowdhury R, Courville KJ, Criqui MH, Cundiff DK, Dabhadkar KC, Dandona L, Davis A, Dayama A, Dharmaratne SD, Ding EL, Durrani AM, Esteghamati A, Farzadfar F, Fay DF, Feigin VL, Flaxman A, Forouzanfar MH, Goto A, Green MA, Gupta R, Hafezi-Nejad N, Hankey GJ, Harewood HC, Havmoeller R, Hay S, Hernandez L, Husseini A, Idrisov BT, Ikeda N, Islami F, Jahangir E, Jassal SK, Jee SH, Jeffreys M, Jonas JB, Kabagambe EK, Khalifa SE, Kengne AP, Khader YS, Khang YH, Kim D, Kimokoti RW, Kinge JM, Kokubo Y, Kosen S, Kwan G, Lai T, Leinsalu M, Li Y, Liang X, Liu S, Logroscino G, Lotufo PA, Lu Y, Ma J, Mainoo NK, Mensah GA, Merriman TR, Mokdad AH, Moschandreas J, Naghavi M, Naheed A, Nand D, Narayan KM, Nelson EL, Neuhouser ML, Nisar MI, Ohkubo T, Oti SO, Pedroza A, Prabhakaran D, Roy N, Sampson U, Seo H, Sepanlou SG, Shibuya K, Shiri R, Shiue I, Singh GM, Singh JA, Skirbekk V, Stapelberg NJ, Sturua L, Sykes BL, Tobias M, Tran BX, Trasande L, Toyoshima H, van de Vijver S, Vasankari TJ, Veerman JL, Velasquez-Melendez G, Vlassov VV, Vollset SE, Vos T, Wang C, Wang X, Weiderpass E, Werdecker A, Wright JL, Yang YC, Yatsuya H, Yoon J, Yoon SJ, Zhao Y, Zhou M, Zhu S, Lopez AD, Murray CJ, Gakidou E. Global, regional, and national prevalence of overweight and obesity in children and adults during 1980-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Aug 30;384(9945):766-81. doi: 10.1016/S0140-6736(14)60460-8. Epub 2014 May 29. PMID 24880830
- [Background] Arterburn D, Gupta A. Comparing the Outcomes of Sleeve Gastrectomy and Roux-en-Y Gastric Bypass for Severe Obesity. JAMA. 2018 Jan 16;319(3):235-237. doi: 10.1001/jama.2017.20449. No abstract available. PMID 29340659
- [Background] Yu EW. Bone metabolism after bariatric surgery. J Bone Miner Res. 2014 Jul;29(7):1507-18. doi: 10.1002/jbmr.2226. PMID 24677277
- [Background] Rousseau C, Jean S, Gamache P, Lebel S, Mac-Way F, Biertho L, Michou L, Gagnon C. Change in fracture risk and fracture pattern after bariatric surgery: nested case-control study. BMJ. 2016 Jul 27;354:i3794. doi: 10.1136/bmj.i3794. PMID 27814663
- [Background] Yu EW, Lee MP, Landon JE, Lindeman KG, Kim SC. Fracture Risk After Bariatric Surgery: Roux-en-Y Gastric Bypass Versus Adjustable Gastric Banding. J Bone Miner Res. 2017 Jun;32(6):1229-1236. doi: 10.1002/jbmr.3101. Epub 2017 Mar 20. PMID 28251687
- [Background] Lalmohamed A, de Vries F, Bazelier MT, Cooper A, van Staa TP, Cooper C, Harvey NC. Risk of fracture after bariatric surgery in the United Kingdom: population based, retrospective cohort study. BMJ. 2012 Aug 3;345:e5085. doi: 10.1136/bmj.e5085. PMID 22867649
- [Background] Lu CW, Chang YK, Chang HH, Kuo CS, Huang CT, Hsu CC, Huang KC. Fracture Risk After Bariatric Surgery: A 12-Year Nationwide Cohort Study. Medicine (Baltimore). 2015 Dec;94(48):e2087. doi: 10.1097/MD.0000000000002087. PMID 26632892
- [Background] Nakamura KM, Haglind EG, Clowes JA, Achenbach SJ, Atkinson EJ, Melton LJ 3rd, Kennel KA. Fracture risk following bariatric surgery: a population-based study. Osteoporos Int. 2014 Jan;25(1):151-8. doi: 10.1007/s00198-013-2463-x. Epub 2013 Aug 3. PMID 23912559
- [Background] Axelsson KF, Werling M, Eliasson B, Szabo E, Naslund I, Wedel H, Lundh D, Lorentzon M. Fracture Risk After Gastric Bypass Surgery: A Retrospective Cohort Study. J Bone Miner Res. 2018 Dec;33(12):2122-2131. doi: 10.1002/jbmr.3553. Epub 2018 Aug 13. PMID 30011091
- [Background] Frederiksen KD, Hanson S, Hansen S, Brixen K, Gram J, Jorgensen NR, Stoving RK. Bone Structural Changes and Estimated Strength After Gastric Bypass Surgery Evaluated by HR-pQCT. Calcif Tissue Int. 2016 Mar;98(3):253-62. doi: 10.1007/s00223-015-0091-5. Epub 2015 Dec 12. PMID 26661530
- [Background] Andersen S, Frederiksen KD, Hansen S, Brixen K, Gram J, Stoving RK. Bone structure and estimated bone strength in obese patients evaluated by high-resolution peripheral quantitative computed tomography. Calcif Tissue Int. 2014 Jul;95(1):19-28. doi: 10.1007/s00223-014-9857-4. Epub 2014 Apr 17. PMID 24736885
- [Background] Shanbhogue VV, Stoving RK, Frederiksen KH, Hanson S, Brixen K, Gram J, Jorgensen NR, Hansen S. Bone structural changes after gastric bypass surgery evaluated by HR-pQCT: a two-year longitudinal study. Eur J Endocrinol. 2017 Jun;176(6):685-693. doi: 10.1530/EJE-17-0014. Epub 2017 Mar 13. PMID 28289103
- [Background] Lindeman KG, Greenblatt LB, Rourke C, Bouxsein ML, Finkelstein JS, Yu EW. Longitudinal 5-Year Evaluation of Bone Density and Microarchitecture After Roux-en-Y Gastric Bypass Surgery. J Clin Endocrinol Metab. 2018 Nov 1;103(11):4104-4112. doi: 10.1210/jc.2018-01496. PMID 30219833
- [Background] Muschitz C, Kocijan R, Marterer C, Nia AR, Muschitz GK, Resch H, Pietschmann P. Sclerostin levels and changes in bone metabolism after bariatric surgery. J Clin Endocrinol Metab. 2015 Mar;100(3):891-901. doi: 10.1210/jc.2014-3367. Epub 2014 Dec 9. PMID 25490275
- [Background] Gagnon C, Schafer AL. Bone Health After Bariatric Surgery. JBMR Plus. 2018 May 1;2(3):121-133. doi: 10.1002/jbm4.10048. eCollection 2018 May. PMID 30283897
- [Background] Schafer AL, Weaver CM, Black DM, Wheeler AL, Chang H, Szefc GV, Stewart L, Rogers SJ, Carter JT, Posselt AM, Shoback DM, Sellmeyer DE. Intestinal Calcium Absorption Decreases Dramatically After Gastric Bypass Surgery Despite Optimization of Vitamin D Status. J Bone Miner Res. 2015 Aug;30(8):1377-85. doi: 10.1002/jbmr.2467. Epub 2015 May 21. PMID 25640580
- [Background] Yu EW, Wewalka M, Ding SA, Simonson DC, Foster K, Holst JJ, Vernon A, Goldfine AB, Halperin F. Effects of Gastric Bypass and Gastric Banding on Bone Remodeling in Obese Patients With Type 2 Diabetes. J Clin Endocrinol Metab. 2016 Feb;101(2):714-22. doi: 10.1210/jc.2015-3437. Epub 2015 Nov 24. PMID 26600045
- [Background] Muschitz C, Kocijan R, Haschka J, Zendeli A, Pirker T, Geiger C, Muller A, Tschinder B, Kocijan A, Marterer C, Nia A, Muschitz GK, Resch H, Pietschmann P. The Impact of Vitamin D, Calcium, Protein Supplementation, and Physical Exercise on Bone Metabolism After Bariatric Surgery: The BABS Study. J Bone Miner Res. 2016 Mar;31(3):672-82. doi: 10.1002/jbmr.2707. Epub 2015 Sep 30. PMID 26350034
- [Background] Mundbjerg LH, Stolberg CR, Bladbjerg EM, Funch-Jensen P, Juhl CB, Gram B. Effects of 6 months supervised physical training on muscle strength and aerobic capacity in patients undergoing Roux-en-Y gastric bypass surgery: a randomized controlled trial. Clin Obes. 2018 Aug;8(4):227-235. doi: 10.1111/cob.12256. Epub 2018 Jun 12. PMID 29896844
- [Background] Frost HM. Bone's mechanostat: a 2003 update. Anat Rec A Discov Mol Cell Evol Biol. 2003 Dec;275(2):1081-101. doi: 10.1002/ar.a.10119. PMID 14613308
- [Background] Tagliaferri C, Wittrant Y, Davicco MJ, Walrand S, Coxam V. Muscle and bone, two interconnected tissues. Ageing Res Rev. 2015 May;21:55-70. doi: 10.1016/j.arr.2015.03.002. Epub 2015 Mar 21. PMID 25804855
- [Background] Black DM, Delmas PD, Eastell R, Reid IR, Boonen S, Cauley JA, Cosman F, Lakatos P, Leung PC, Man Z, Mautalen C, Mesenbrink P, Hu H, Caminis J, Tong K, Rosario-Jansen T, Krasnow J, Hue TF, Sellmeyer D, Eriksen EF, Cummings SR; HORIZON Pivotal Fracture Trial. Once-yearly zoledronic acid for treatment of postmenopausal osteoporosis. N Engl J Med. 2007 May 3;356(18):1809-22. doi: 10.1056/NEJMoa067312. PMID 17476007
- [Background] Boonen S, Reginster JY, Kaufman JM, Lippuner K, Zanchetta J, Langdahl B, Rizzoli R, Lipschitz S, Dimai HP, Witvrouw R, Eriksen E, Brixen K, Russo L, Claessens F, Papanastasiou P, Antunez O, Su G, Bucci-Rechtweg C, Hruska J, Incera E, Vanderschueren D, Orwoll E. Fracture risk and zoledronic acid therapy in men with osteoporosis. N Engl J Med. 2012 Nov 1;367(18):1714-23. doi: 10.1056/NEJMoa1204061. PMID 23113482
- [Background] Deas CM, Murphy P, Iranikhah M, Freeman MK. Retained Skeletal Effects of Zoledronic Acid Following Discontinuation of Treatment: A Review of the Literature. Consult Pharm. 2017 Mar 1;32(3):144-155. doi: 10.4140/TCP.n.2017.144. PMID 28270269
- [Background] Watanabe R, Fujita N, Takeda S, Sato Y, Kobayashi T, Morita M, Oike T, Miyamoto K, Matsumoto Y, Matsumoto M, Nakamura M, Miyamoto T. Ibandronate concomitantly blocks immobilization-induced bone and muscle atrophy. Biochem Biophys Res Commun. 2016 Nov 25;480(4):662-668. doi: 10.1016/j.bbrc.2016.10.112. Epub 2016 Oct 27. PMID 27983979
- [Background] Borsheim E, Herndon DN, Hawkins HK, Suman OE, Cotter M, Klein GL. Pamidronate attenuates muscle loss after pediatric burn injury. J Bone Miner Res. 2014 Jun;29(6):1369-72. doi: 10.1002/jbmr.2162. PMID 24347438
- [Derived] Gam S, Hermann AP, Juhl CB, Hansen SG, Gram B. Effect of Zoledronic Acid on Skeletal Muscle After Bariatric Surgery: A Secondary Analysis From a Randomized Controlled Trial. Obesity (Silver Spring). 2026 Jan;34(1):76-87. doi: 10.1002/oby.70062. Epub 2025 Nov 2. PMID 41177144
- [Derived] Gam S, Gram B, Juhl CB, Hermann AP, Hansen SG. Zoledronic Acid for prevention of bone and muscle loss after BAriatric Surgery (ZABAS)-a study protocol for a randomized controlled trial. Trials. 2022 Oct 8;23(1):861. doi: 10.1186/s13063-022-06766-z. PMID 36209245